CLINICAL TRIAL: NCT02001675
Title: Comparison of Both Metabolic and Functional Effects Induced by Two Neuromuscular Electrical Stimulation Protocols: A Comprehensive Approach Using Magnetic Resonance Imaging and Spectroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A01265-38; 2012-32 (Other: AP HM)
Record Dates: First submitted 2012-12-21; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Neuromuscular electrical stimulation (NMES)
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volunteer healthy (Experimental)
  Interventions: Device: magnetic resonance imaging (MRI); Device: 31-phosphorous magnetic resonance spectroscopy (MRS-P31)

INTERVENTIONS:
Device: magnetic resonance imaging (MRI)
Device: 31-phosphorous magnetic resonance spectroscopy (MRS-P31)

SUMMARY:
Neuromuscular electrical stimulation (NMES) has emerged as a suitable tool for restoring, maintaining and/or enhancing muscular performance. From a practical point of view, NMES can elicit contractions either by direct activation of motor axons (i.e. peripheral mechanism) or by the recruitment of motoneurons in the spinal cord through the depolarization of sensory axons (central mechanism). It is noteworthy that NMES parameters widely affect the balance between transmission along these two pathways. Conventional NMES is usually delivered using short pulse duration (0.05-0.4 ms), low stimulation frequency (15-40 Hz) and high stimulus intensities so that the large antidromic volley in motor axons ensures that the evoked contraction will be driven largely by the direct depolarization of motor axons beneath the stimulation site with no or little involvement of central nervous system. On the contrary, when NMES is delivered using wide pulse widths (1 ms) and high frequency (up to 100 Hz) (WP-HF NMES), a portion of the evoked contraction arises from a central mechanism and the corresponding force (recently referred to as "extra force") is significantly (three times) larger than the conventional NMES-induced force. This extra force is supposed to represent the central contribution from the recruitment of spinal motoneurons by the evoked afferent volley given that no additional force was observed during a complete anesthetic block of the nerve proximal to the stimulation site. Despite the obvious differences in terms of activation of the neuromuscular system between conventional and WP-HF NMES, the functional, metabolic and cortical responses associated to both protocols remain to be determined

DETAILED DESCRIPTION:
The main goal of the project will be to characterize the evoked-force profile during conventional and WP-HF NMES.

The secondary purpose will be to i) investigate the anatomic and metabolic responses of the human calf muscle following both NMES protocols by using magnetic resonance imaging (MRI) and 31-phosphorous magnetic resonance spectroscopy (MRS-P31), ii) study the cortical responses for both conditions of stimulation by means of functional MRI (f-MRI).

ELIGIBILITY:
Inclusion Criteria:

* age included between 18 and 45 years
* The volunteers will have to benefit from a social security cover.
* The selected subjects will have to be unhurt of any general disease, psychiatric disorders and any infectious, inflammatory, tumoral, vascular, degenerative or traumatic pathology.

They will have to follow no chronic treatment and will have to be unhurt of any history of alcoholism or drug addiction.

Exclusion Criteria:

* Usual contraindications for an examination MRI.

So, will not be included, the subjects:

* suffering from claustrophobia,
* having stimulating one cardiac, carriers of a system Holter,
* carriers of hook(staple) (clip) surgical metallic,
* Carriers of a prosthesis or a metallic implant (or quite different metallic foreign bodies),
* carriers of a prosthesis dental (device),
* carriers of a hearing aid,
* carriers of an insulin pump,
* having been hurt by pieces of shrapnel or lead,
* Having had a dislocation, a fracture or a recent surgical operation (less than 6 months before the inclusion),
* Having followed a treatment(processing) with anti-inflammatory drugs during the last 3 months, having followed a treatment(processing) with amino acids during 3

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
RMI | 36 months
  Assessment of muscle function or brain

CONTACTS AND LOCATIONS:
Overall Officials: michele DAMON, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France